CLINICAL TRIAL: NCT03422315
Title: Population Pharmacokinetics and Clinical Individual Dosage Regimen of Propofoll Injection in Adult Patients With General Anesthesia
Brief Title: Population Pharmacokinetics and Clinical Individual Dosage Regimen of Propofoll Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongyuan Xu (Other)
Responsible Party: Sponsor-Investigator, Zhongyuan Xu, Director of GCP Office, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C1033453
Record Dates: First submitted 2017-06-08; First posted 2018-02-05 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-03

CONDITIONS: General Anesthesia
Keywords: Propofol; Population pharmacokinetics; Individualized administration
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- External control (Experimental): propofol;injection;2mg/kg;single-dose
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — injection;2mg/kg;single-dose

SUMMARY:
Propofol is a widely used sedative anesthetic, but there are large individual differences, which making different patients with different sensitivity to propofol. The aim of this study was to analyze the effects of age, height, body weight, Drinking, metabolic enzymes CYP2B6 and UGT1A9 on Pharmacological effects and pharmacokinetics of propofol, and to provide a reasonable reference for clinical anesthesia patients and evidence for individual dosage regimens.

DETAILED DESCRIPTION:
Propofol is a widely used sedative anesthetic, but there are large individual differences, which making different patients with different sensitivity to propofol. In recent years, the concept of individualized administration came into being.Individual administration refers to according to the condition of patients,the drug's safety and efficacy, and pharmacokinetics, pharmacodynamics and clinical response ,then gives different dosing regimens for individual patients and promotes the development of rational drug use. Different people have differences metabolism of propofol, reported in the literature, genetic polymorphism, demographic characteristics, combined with drug and other variability factors, all of them will affect the pharmacokinetics and pharmacodynamics of propofol.The aim of this study was to analyze the effects of age, height, body weight, Drinking, metabolic enzymes CYP2B6 and UGT1A9 on Pharmacological effects and pharmacokinetics of propofol, and to provide a reasonable reference for clinical anesthesia patients and evidence for individual dosage regimens.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-60 years (including those aged 18 and 60) who underwent gastrointestinal endoscopy;
* weight should not be less than (≥) 50kg, not more than (≤) 80kg. Body mass index (BMI) = body weight kg / [(height m) 2], in the normal range of 19 to 25;
* American Society of Anesthesiologists (ASA) grading (Appendix I): I or II;
* no heart, liver, lung, kidney, digestive tract, nervous system, mental disorders and other medical history, no blood and metabolic diseases and other medical history, no potential difficulties airway and special past history,
* blood, urine, stool routine, liver and kidney function, blood lipids, ECG, chest X-ray and blood pressure normal, or abnormal but no clinical significance, the researchers believe that can be grouped.
* agree and sign informed consent.

Exclusion Criteria:

* important organs have primary disease;
* persons with mental or physical disabilities;
* those suffering from neurological or mental illness, a history of epilepsy;
* patients with cardiovascular or respiratory insufficiency and hypovolemia;
* obese or those with dyslipidemia;
* hereditary acute porphyria;
* infections, especially those with respiratory and central infections;
* language exchange barriers;
* suspected or indeed a history of alcohol, drug abuse; especially long-term use of non-steroidal anti-inflammatory drugs, opioids, tranquilizers;
* allergies, if the history of drugs or food allergies; or known to propofol, soybeans, peanuts, coconut oil allergy;
* smoking history (smoking ≥ 5 per day);
* 2 weeks before the trial had used all kinds of Chinese and Western medicine;
* the last 3 months of blood donors and test blood donors;
* other circumstances that the researcher thinks can not be grouped (eg, frail, etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2018-09-03 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
BIS | 210min
  bispectral index monitoring

CONTACTS AND LOCATIONS:
Overall Officials: zhongyuan xu, Ph.D., Study Director — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital，Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kansaku F, Kumai T, Sasaki K, Yokozuka M, Shimizu M, Tateda T, Murayama N, Kobayashi S, Yamazaki H. Individual differences in pharmacokinetics and pharmacodynamics of anesthetic agent propofol with regard to CYP2B6 and UGT1A9 genotype and patient age. Drug Metab Pharmacokinet. 2011;26(5):532-7. doi: 10.2133/dmpk.dmpk-11-rg-039. Epub 2011 Aug 23. PMID 21869535
- [Background] Bernard O, Guillemette C. The main role of UGT1A9 in the hepatic metabolism of mycophenolic acid and the effects of naturally occurring variants. Drug Metab Dispos. 2004 Aug;32(8):775-8. doi: 10.1124/dmd.32.8.775. PMID 15258099
- [Background] Takahashi H, Maruo Y, Mori A, Iwai M, Sato H, Takeuchi Y. Effect of D256N and Y483D on propofol glucuronidation by human uridine 5'-diphosphate glucuronosyltransferase (UGT1A9). Basic Clin Pharmacol Toxicol. 2008 Aug;103(2):131-6. doi: 10.1111/j.1742-7843.2008.00247.x. PMID 18816295
- [Background] Khan MS, Zetterlund EL, Green H, Oscarsson A, Zackrisson AL, Svanborg E, Lindholm ML, Persson H, Eintrei C. Pharmacogenetics, plasma concentrations, clinical signs and EEG during propofol treatment. Basic Clin Pharmacol Toxicol. 2014 Dec;115(6):565-70. doi: 10.1111/bcpt.12277. Epub 2014 Jul 19. PMID 24891132